CLINICAL TRIAL: NCT02280226
Title: Evaluating the Influence of Apnea on Heart Function With Strain Analysis and Measurement of Fibrosis Derived From T1-mapping Using Cardiac Magnetic Resonance Imaging (MRI).
Brief Title: Evaluating the Influence of Apnea on Cardiac Function Using Cardiac Magnetic Resonance Imaging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Jonas Doerner, MD, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UBonn-MRI-heart-14
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Physiological Changes in Deliberate Apnea
MeSH Terms: interventions — Magnetic Resonance Imaging

ARMS (1):
- Deliberate Apnea Group (Experimental): Subjects undergo maximum apnea.
  Interventions: Device: magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: magnetic resonance imaging (MRI)

SUMMARY:
Former studies revealed a distinct pattern of changes in circulation during deliberate apnea. Blood pressure rises significantly often accompanied by bradycardia. Further studies confirmed a massive increase of total vascular resistance as it also happens in shock to maintain perfusion of heart, lung and brain. This study is to determine the exact alterations of the cardiac function during this reaction, show the redistribution of blood volume in apnea and evaluate possible longterm effects on the central nervous system caused by repeated apnea via magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Being able to hold breath deliberately at least 4,5 minutes

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

REFERENCES:
- [Derived] Eichhorn L, Doerner J, Luetkens JA, Lunkenheimer JM, Dolscheid-Pommerich RC, Erdfelder F, Fimmers R, Nadal J, Stoffel-Wagner B, Schild HH, Hoeft A, Zur B, Naehle CP. Cardiovascular magnetic resonance assessment of acute cardiovascular effects of voluntary apnoea in elite divers. J Cardiovasc Magn Reson. 2018 Jun 18;20(1):40. doi: 10.1186/s12968-018-0455-x. PMID 29909774

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deliberate Apnea Group
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Deliberate Apnea Group: Subjects undergo maximum apnea.
  magnetic resonance imaging (MRI)
Arm/Group | Deliberate Apnea Group
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 16
  Switzerland | 1

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Function: Duration of Apnea
Description: Alteration of cardiac function in subjects undergoing maximum apnea.
Time Frame: every minute under apnea (from 0 up to 9 minutes and rest) depending on personal best with a mean of 5 measurements
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Deliberate Apnea Group
Number analyzed (Participants) | 17
sec | 483 (582)

2. Primary Outcome: Mean Blood Flow Measurement Under Apnea Using MRI
Description: Blood flow pattern in subjects undergoing maximum apnea.
Time Frame: Every minute under apnea (from 0 up to 9 minutes and rest) depending on personal best with a mean of 5 measurements
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Deliberate Apnea Group
Number analyzed (Participants) | 17
ml/s | 82 (27)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- Deliberate Apnea Group: Subjects undergo maximum apnea and magnetic resonance imaging (MRI) was performed.
Arm/Group | Deliberate Apnea Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No